CLINICAL TRIAL: NCT02297048
Title: Monocentric STUDY, Randomised Double Blinded (Healthy Subjects, or Transversal (Patients With Gitelman Syndrome)
Acronym: DEPROGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P120906
Record Dates: First submitted 2014-10-29; First posted 2014-11-21 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Gitelman Syndrome; Potassium Depletion
Keywords: Potassium intake; Progesterone; steroidogenesis; RU486; Synachtene test
MeSH Terms: conditions — Gitelman Syndrome; Hypokalemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RU 486 (mifepristone) (Experimental): Subjects will receive 400 mg once a day of RU486
  Interventions: Dietary Supplement: Potassium depletion
- Placebo (Placebo Comparator): Subjects will receive placebo once a day
  Interventions: Dietary Supplement: Potassium depletion

INTERVENTIONS:
Dietary Supplement: Potassium depletion — Healthy subjects will be submitted twice at 15-30 day interval, to a low potassium diet (20mmol/day)

SUMMARY:
Progesterone is needed to permit adaptation of the kidney to limit potassium loss in the urines. The investigators wonder whether progesterone or other adrenal hormon play the same role. The investigators will investigate surrenal hormone production in healthy subjects under a 7-day potassium depleted diet and in patients chronically hypokalaemic due to a renal loss of potassium.

DETAILED DESCRIPTION:
The investigators will study the adaptation of steroidogenesis to potassium depletion in healthy volunteer, and the role of progesterone in renal adaptation to potassium depletion. Practically, healthy volunteers will be submitted twice to two periods of normal Na+/ high K+ diet (control period) followed by a normal Na+/ low K+ diet sustained by a pharmacological treatment with Kayexalate (K+-depleted condition). The subjects will be treated with either RU486 or a placebo, according to a randomization. The adrenal response will be evaluated after stimulation by Synacthen at baseline and at the end of each experimental period. A Synacthen test will be also done in 10 patients suffering of chronic hypokalemia linked to a hereditary tubulopathy inducing renal K+ leak called Gitelman syndrome and their plasma steroid profile will be established.

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* Caucasian male subject
* 18-35 yrs-old
* BMI between 18 and 30 Kg/m2
* Normal biological pattern (sodium, potassium, eGFR >60mL/min/1.73 m2, SGOT and SGPT < 2.5 normal value)
* Non smoker subjects or less than 5 cigarettes a day
* No drug abuse
* No active viral B or C hepatitis, no positive HIV serology
* No treatment except paracetamol
* Normal EKG
* Inform consent given
* Affiliation to French Medicare assurance

Inclusion Criteria for patients :

* 18-75 Years old subjects
* genetically proven Gitelman syndrome
* Normal EKG
* Inform consent given
* Affiliation to French Medicare assurance

Non inclusion Criteria for healthy subjects:

* History of cardiac arrythmia or abnormal EKG
* Recent or chronic diarrhea
* Spontaneous low potassium intakes
* Biological abnormality : SGOT or SGPT > 2.5 N, fasting hyperglycemia (> 6.5 mmol/l, anemia (hemoglobin< 12g/dL)
* Single or functionally solitary kidney
* Any severe allergies, or allergic history to any drug.
* Predicted Difficulty monitoring and compliance.
* Blood donation for less than 2 months.
* Persons directly involved in the implementation of the Protocol.
* Person in exclusion period in biomedical research.
* Protected Person (person under guardianship, deprived of liberty, ...).
* Taking medication in the previous 7 days (except paracetamol).
* Chronic adrenal insufficiency.
* Known allergy to any of the excipients of the RU 486 (colloidal anhydrous silica, maize starch, povidone, microcrystalline cellulose, magnesium stearate).
* Severe asthma not controlled by treatment.
* Porphyria hereditary.

Non inclusion Criteria for Gitelman patients:

* People that did not give their consent or unable to understand the protocol.
* Anemia (Hg <10 g / dL).
* Clinically significant abnormality on the EKG.
* Any severe allergies, or allergic history to any drug.
* Treatment with corticosteroids.
* Patient in exclusion period in biomedical research.
* Protected Person (patient trust, deprived of liberty, ...)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effect of potassium depletion on plasma progesterone (Change from Baseline of progesterone) | Day 1 and Day 8 of placebo period of treatment (healthy subjects) or once (Gitelman patients)
  Healthy subjects : Change from Baseline of progesterone in response to synacthen at day 8 in subject treated by placebo.
  Patients with Gitelman syndrome: Change from Baseline of progesterone in response to synacthen

SECONDARY OUTCOMES:
effect of RU 486 on renal adaptation to potassium depletion (Plasma potassium and kaliuresis will be monitored ) | Day 1 and day 8 of each period of treatment
  Plasma potassium and kaliuresis will be monitored during the 7-days potassium depletion in subjects treated by RU486 or placebo, according randomization
Effect of potassium depletion on pulse pressure velocity (Pulse wave velocity and central blood pressure) | At Day 1 and Day 8 of each period of treatment
  Pulse wave velocity and central blood pressure are measured before and after 7 days of potassium deprivated diet.
Effect of potassium depletion on plasma progesterone under RU486 (Change from Baseline of progesterone) | Day 1 and Day 8 of placebo period of treatment (healthy subjects) or once (Gitelman patients)
  Healthy subjects : Change from Baseline of progesterone in response to synacthen at day 8 in subject treated by RU486.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Blanchard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- European George Pompidou Hospital, Paris, France

REFERENCES:
- [Background] Elabida B, Edwards A, Salhi A, Azroyan A, Fodstad H, Meneton P, Doucet A, Bloch-Faure M, Crambert G. Chronic potassium depletion increases adrenal progesterone production that is necessary for efficient renal retention of potassium. Kidney Int. 2011 Aug;80(3):256-62. doi: 10.1038/ki.2011.15. Epub 2011 Feb 16. PMID 21326170
- [Derived] Blanchard A, Brailly Tabard S, Lamaziere A, Bergerot D, Zhygalina V, Lorthioir A, Jacques A, Hourton D, Azizi M, Crambert G. Adrenal adaptation in potassium-depleted men: role of progesterone? Nephrol Dial Transplant. 2020 Nov 1;35(11):1901-1908. doi: 10.1093/ndt/gfz135. PMID 31369102